CLINICAL TRIAL: NCT06110403
Title: Impact of Inhaled BGF 160 on Complexity and Variability of Tidal Breathing and Oscillatory Mechanics in Stable COPD Patient
Brief Title: Impact of Long-acting Bronchodilator- -Corticoid Inhaled Therapy on Ventilation, Lung Function and Breathlessness
Acronym: VARI-OSCIL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022_0422; 2022-003784-15 (EudraCT Number)
Record Dates: First submitted 2023-02-21; First posted 2023-10-31 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Copd
Keywords: COPD; bronchodilator; ventilatory mode; variability; forced oscillations; spirometry; plethysmography; dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Symptomatic COPD patients in stable condition treated with BGF 160 (Trixéo Aerosphere®), a combination of budesonide, formoterol and glycopyrronium in a metered dose inhaler, taken twice a day
  Interventions: Drug: TRIXEO AEROSPHERE

INTERVENTIONS:
Drug: TRIXEO AEROSPHERE — BGF 160 (Breztri Aerosphere™ in USA, Trixeo™ in France) Inhalation aerosol: pressurized metered dose inhaler containing a combination of budesonide (160 mcg), glycopyrrolate (9 mcg) and formoterol fumarate (4.8 mcg) as an inhalation aerosol. Oral inhalation: 2 inhalations of BGF 160 twice daily for 30 days.

SUMMARY:
Multicentre, prospective, non-randomised, single-arm, open label, mechanistic study to investigate the mechanism of action of BGF 160 on ventilation pattern complexity and variability

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed informed consent prior to any study specific procedure
* Female or male subjects aged 40-75 years inclusive at the time of enrolment (Visit 1)
* Documented history of COPD with a post-bronchodilator FEV1/FVC <0.70 and a post-bronchodilator 30 % < FEV1 <70% of predicted normal value (according to ERS 1993 reference values for spirometry ) at screening
* Smoking history > 10 pack-years
* Baseline significant dyspnea with a mMRC ≥ 2

Exclusion Criteria:

* History or current diagnosis of asthma or ACOS (asthma-COPD overlap syndrome)
* Respiratory infection or COPD exacerbation within 6 weeks (2 months if it resulted in hospitalization) prior to screening
* Clinically significant or relevant cardiovascular conditions, laboratory tests, electrocardiogram (ECG) parameters:

  * Unstable angina/acute coronary syndrome, or Coronary Artery Bypass Grafting (CABG), Percutaneous Coronary Intervention (PCI) or myocardial infarction within the past 6 months.
  * Congestive heart failure New York Heart Association (NYHA) class III/IV.
  * Structural heart disease (hypertrophic cardiomyopathy, significant valvular disease).
  * Paroxysmal (within the past 6 months) or symptomatic chronic cardiac tachyarrhythmia.
  * Left bundle branch or high-degree AV block (second degree AV block type 2 and third degree AV block) unless the patient has a pacemaker.
  * Sinus node dysfunction with pauses.
  * Ventricular pre-excitation and/or Wolff-Parkinson-White syndrome.
  * QTcF interval >470 msec (QT interval corrected using Fridericia's formula; QTcF=QT/[RR1/3]).
  * Any other ECG abnormality deemed clinically significant by the Investigator.
  * Bradycardia with ventricular rate < 45 bpm.
  * Uncontrolled hypertension (> 165/95 mmHg).
* Clinically relevant respiratory conditions (other than COPD)
* Severe renal impairment eGFR < 30
* Hepatic impairment
* Narrow-angle glaucoma that, in the opinion of the Investigator, has not been adequately treated.
* Symptomatic prostatic hypertrophy or bladder neck obstruction/urinary retention that is clinically significant
* Patients not able to perform IOS, spirometry, plethysmography, or VT acquisition (10 min)
* Any contraindication to LABA or LAMA drugs or to Inhaled corticosteroids
* Pregnancy or breastfeeding
* Woman of childbearing age without effective contraception
* Any type of cancer within 5 years
* Patients under guardianship
* Refuse or incapacity to give an informed consent
* Absence of social insurance

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
change in ventilation pattern complexity and variability | between V2 baseline (pre-treatment) and V3 peak (2 hours (+/-30minutes) post dose at one month)
  * Noise limit: %
  * Lyapounov component: bits/iteration no combination possible

SECONDARY OUTCOMES:
Change impulse oscillometry or forced oscillation: resistances at 5Hz, reactance at 5Hz | between V2 base (pre-treatment) and V3 peak (2 hours (+/-30minutes) post dose
  resistance and reactance: kPa/L/s
Changes in FEV1 (spirometry) | between V2 base (pre-treatment) and V3 peak (2 hours (+/-30minutes) post dose
Change Plethysmographic Functional residual capacity (FRC) | between V2 base (pre-treatment) and V3 peak (2 hours (+/-30minutes) post dose
Changes measurement for noise limit, respiratory frequency, volume, largest Lyapounov component, resistances at 5Hz, reactance at 5Hz, FEV1and FRC versus TDI at V3 | between V2 base measurement (pre-treatment) and V3 peak (2 hours (+/-30min)
  TDI at V3 (in term of continuous variable and in term of binary variable "responder/non responder"; a response is defined by a change in TDI ≥ +1 between baseline and V3)
Baseline dyspnea index ( BDI) | before administration of BGF 160 (at V2 base (pre-treatment)) and after administration (at V3 peak (2 hours (+/-30minutes) at one month)
Transition dyspnea index (TDI) | before administration of BGF 160 (at V2 base (pre-treatment)) and after administration (at V3 peak (2 hours (+/-30minutes) at one month)
Modified dyspnea profile ( MDP) | before administration of BGF 160 (at V2 base (pre-treatment)) and after administration (at V3 peak (2 hours (+/-30minutes) at one month)
CAT score : COPD assessment test, | before administration of BGF 160 (at V2 base (pre-treatment)) and after administration (at V3 peak (2 hours (+/-30minutes at one month)
  range 0 to 40, 40 meaning the worst condition
Likert scale for dyspnea and general health | before administration of BGF 160 (at V2 base (pre-treatment)) and after administration (at V3 peak (2 hours (+/-30minutes) at one month)
  Likert scale change in dyspnea : - 3 to + 3, + 3 maximal improvement, -3 maximal deterioration Likert scale change in general health : - 3 to + 3, + 3 maximal improvement, -3 maximal deterioration

CONTACTS AND LOCATIONS:
Overall Officials: Thierry PEREZ, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHU de Lille, Lille, France